CLINICAL TRIAL: NCT01274234
Title: Evaluation of Neointimal Healing of Endothelial Progenitor Cell Capturing Sirolimus-Eluting (COMBO) Stent by Optical Coherence Tomography: the EGO-COMBO Pilot Study
Brief Title: OCT Evaluation of Healing of COMBO Stent
Acronym: EGO-COMBO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prof. Stephen Lee (Other)
Responsible Party: Sponsor-Investigator, Prof. Stephen Lee, Professor and Chief, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UW 10-342 (IRB HKU)
Record Dates: First submitted 2010-12-28; First posted 2011-01-11 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Coronary Restenosis; Coronary Thrombosis
Keywords: EPC capturing sirolimus eluting COMBO stent; Optical coherence tomography (OCT); Early neointimal healing and stent coverage; Late neointimal thickness, neointimal area, and lumen loss
MeSH Terms: conditions — Coronary Restenosis; Coronary Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- COMBO Stent (Experimental): COMBO Stent
  Interventions: Device: COMBO Stent (OrbusNeich Medical, Fort Lauderdale, Florida)

INTERVENTIONS:
Device: COMBO Stent (OrbusNeich Medical, Fort Lauderdale, Florida) — The COMBO Stent is a hybrid version of the GENOUS Stent. Upon implantation to the coronary artery, the stent will deliver a drug (sirolimus) to the wall of the treated segment to suppress neointimal growth, in addition to the anti-CD34 antibody coating which will in theory attract circulatory endothelial progenitor cells to hasten endothelialization and promote healing of the stented segment, and thereby may reduce late stent thrombosis.
  Other Names: COMBO Stent

SUMMARY:
All subjects requiring percutaneous coronary intervention (PCI) and stenting are eligible to participate in the study. Restudy coronary angiogram with Optical Coherence Tomography (OCT) would be performed between 1 to 5 months at the time of a staged PCI procedure (for remaining coronary disease) or as clinically indicated, and then at 9 months. At the time of the 9-month restudy (a proper time window for drug eluting stent to develop into restenosis should it occur), any new disease detected or restenosis will be treated. The reported incidence of drug eluting stent restenosis is around 10% in simple lesions and is expected to be higher in diabetic patients, long lesions and multi-vessel diseases; a restudy at 9 months actually confers better protection to the patients with advanced disease and any restenosis can be treated timely. All data on clinical events and progress will be monitored and regular follow-ups will be carried out.

DETAILED DESCRIPTION:
The GENOUS Stent (the EPC Capturing R-stent, OrbusNeich Medical Inc., Fort Lauderdale, FL) is commercially available and has been extensively used in standard coronary intervention procedures treating >200 patients with critical coronary stenoses at Queen Mary Hospital. The COMBO Stent (OrbusNeich Medical Inc., Fort Lauderdale, FL) is a hybrid version of the GENOUS Stent with an abluminal sirolimus coating, and is currently under the investigational use for clinical research in the REMEDEE Study; over 20 patients have been treated and all remained in good condition since the treatment.

The GENOUS Stent is a bio-engineered 316L stainless steel coronary stent with a biocompatible circumferential coating of anti-CD34 antibody, and will bind to and therefore capture the circulatory endothelial progenitor cells (EPC) which have CD34 antigen on the surface. Immobilization of EPCs on the stent surface will encourage differentiation and proliferation of the EPCs into endothelial and neointimal layer. Animal model has demonstrated that a functional endothelial layer could be formed as soon as 24 to 48 hours after GENOUS stent implantation (1). The HEALING-FIM registry has shown that GENOUS stent is clinically safe and effective in the treatment of coronary stenosis (2). Recent reports have further confirmed its efficacy in patients with acute coronary syndrome requiring urgent revascularization (3,4).

The COMBO Stent is a hybrid version of the GENOUS Stent, with an additional abluminal, drug eluting sirolimus coating, targeted to reduce excessive neointima formation, while maintaining the EPC capturing capacity and therefore continue to promote healing after stent injury. The hybrid function of these two technologies in this new COMBO stent is expected to produce better clinical results in terms of accelerated healing, less stent thrombosis and less restenosis; these are being investigated in the current REMEDEE Study.

Animal study has shown the COMBO Stent promotes endothelialization and reduces neointima formation, as assessed by both optical coherence tomography (OCT) and histopathology (5). Even though COMBO Stents have been used and found to be safe in over 180 patients world-wide and in about 30 patients at Queen Mary Hospital under the REMEDEE Study Protocol, such benefits of "early" endothelial coverage as assessed by OCT has never been fully documented in human subjects.

The current EGO-COMBO study protocol is designed based on the approved protocols of the ongoing REMEDEE Study (IRB: UW 09-384) and the EGO Study (IRB: UW 10-256); both are still active in this Hospital. In the multi-center REMEDEE Study, the COMBO stent is compared to the TAXUS stent (Boston Scientific) in patients with coronary artery disease requiring stent implantation, looking at the 9 months late loss results. This EGO-COMBO Study is different from the REMEDEE Study and focuses mainly on the very early time frames assessing the degree of early neointimal healing (enhanced endothelialization) between 2nd to 5th months, and the subsequent neointimal proliferation at 9 months after the COMBO Stent implantation, as assessed by the very high resolution of the frequency domain optical coherence tomography (OCT) used in the existing EGO study. This is a single centre, non-randomized, open-label study.

Intracoronary frequency domain optical coherence tomography (FD-OCT) is a simple catheter-based imaging technique using optic fibre to achieve very detailed assessment (resolution down to 10 microns) of the stents, in terms of stent apposition, early neointimal coverage (enhanced endothelialization) and late stent neointimal growth (restenosis). It is performed as part of the routine cardiac catheterization procedure and provides high-resolution cross sectional images of the coronary arteries. OCT has been shown to be safe in clinical practice (6, 7). The LightLab C7XR OCT System (Frequency Domain OCT) is a commercially available product with CE Mark and FDA approval, and is being used in our EGO Study. The Dragonfly OCT catheter used is a non-occlusive optic fibre which is extremely small and flexible, and will pose absolutely no additional risk to the patient under treatment, other than those inherent risks of a standard angioplasty procedure.

In this prospective, pilot study, OCT is used to image the COMBO Stent after implantation to evaluate both the early healing (stent apposition, neointimal coverage) and late lumen loss (neo-intimal thickness and neo-intimal area). Clinical outcomes will also be monitored as secondary end points. The OCT analyses will be performed by an USA based core laboratory, which is blinded from the time frame of the OCT pullbacks and the clinical details.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 18-85 years old,
* patient with coronary stenosis requiring percutaneous coronary intervention without contraindications to implantation of drug eluting stents
* patient who consents to receive follow-up coronary angiogram and OCT examination.

Exclusion Criteria:

- patient who refuses to consent to follow-up coronary angiogram or OCT examination.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Primary end-point: OCT findings on percentage stent strut coverage in the 2nd to the 5th months (4 monthly groups). | On 2nd, 3rd, 4th, and 5th months
  Primary end-point: OCT findings on percentage stent strut coverage, malapposition, and neointimal thickness in the 2nd to the 5th months (4 monthly groups).

SECONDARY OUTCOMES:
OCT findings on late loss (neointimal thickness and neointimal area) at 9 months restudy. | 9 months
  OCT findings on late loss (neointimal thickness, neointimal area, percentage plaque volume, lumen area, and late loss in lumen area) at 9 months restudy.
Major Adverse Cardiac Events | Initial OCT follow up, 9 months follow up and one year follow up
  Major Adverse Cardiac Events (MACE) which defined as:
  1. Death from all cause including cardiac death
  2. Any Myocardial Infarction (Q wave and non Q-wave)
  Elevation of post-procedure CK levels to greater 2 times normal without new Q waves is considered a non Q-wave MI.
  Development of new, pathological Q waves in 2 or more contiguous leads,as assessed by the investigator and confirmed by the Clinical Endpoint Committee and elevation of cardiac enzymes. In the absence of ECG data the CEC may adjudicate Q wave MI based on the clinical scenario and appropriate cardiac enzyme data.
Major Adverse Cardiac Events | Initial OCT follow up, 9 months OCT follow up and one year follow up
  3. Target Lesion Revascularization requiring repeat PCI or CABG to the target lesion. Clinically driven Revascularization at the target lesion associated with positive functional ischemia study or ischemic symptoms AND an angiographic minimal lumen diameter stenosis ≥50% by QCA, or revascularization of a target lesion with diameter stenosis ≥ 70% by QCA without either angina or a positive functional study.
Any Stent Thrombosis according the Academic Research Consortium | Initial OCT follow up, 9 months OCT follow up and one year follow up
Stroke | Initial OCT follow up, 9 months OCT follow up and one year follow up
  Stroke defined as sudden onset of vertigo, numbness, dysphasia, weakness, visual field defects, dysarthria or other focal neurological deficits due to vascular lesions of the brain such as hemorrhage, embolism, thrombosis, or rupturing aneurysm, that persists more than 24 hours.
Bleeding complication | Initial OCT follow up, 9 months OCT follow up and one year follow up
  Bleeding complication defined as a procedure related hemorrhagic event that requires a transfusion or surgical repair. These may include a hematoma requiring treatment of retroperitoneal bleed.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lee, MD FRCP FACC, Principal Investigator — Queen Mary Hospital, The Unversity of Hong Kong
Locations (1):
- Division of Cardiology, Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Result] Aoki J, Serruys PW, van Beusekom H, Ong AT, McFadden EP, Sianos G, van der Giessen WJ, Regar E, de Feyter PJ, Davis HR, Rowland S, Kutryk MJ. Endothelial progenitor cell capture by stents coated with antibody against CD34: the HEALING-FIM (Healthy Endothelial Accelerated Lining Inhibits Neointimal Growth-First In Man) Registry. J Am Coll Cardiol. 2005 May 17;45(10):1574-9. doi: 10.1016/j.jacc.2005.01.048. PMID 15893169
- [Result] Co M, Tay E, Lee CH, Poh KK, Low A, Lim J, Lim IH, Lim YT, Tan HC. Use of endothelial progenitor cell capture stent (Genous Bio-Engineered R Stent) during primary percutaneous coronary intervention in acute myocardial infarction: intermediate- to long-term clinical follow-up. Am Heart J. 2008 Jan;155(1):128-32. doi: 10.1016/j.ahj.2007.08.031. Epub 2007 Nov 26. PMID 18082503
- [Result] Miglionico M, Patti G, D'Ambrosio A, Di Sciascio G. Percutaneous coronary intervention utilizing a new endothelial progenitor cells antibody-coated stent: a prospective single-center registry in high-risk patients. Catheter Cardiovasc Interv. 2008 Apr 1;71(5):600-4. doi: 10.1002/ccd.21437. PMID 18360849
- [Result] Granada JF, Inami S, Aboodi MS, Tellez A, Milewski K, Wallace-Bradley D, Parker S, Rowland S, Nakazawa G, Vorpahl M, Kolodgie FD, Kaluza GL, Leon MB, Virmani R. Development of a novel prohealing stent designed to deliver sirolimus from a biodegradable abluminal matrix. Circ Cardiovasc Interv. 2010 Jun 1;3(3):257-66. doi: 10.1161/CIRCINTERVENTIONS.109.919936. Epub 2010 May 4. PMID 20442358
- [Result] Yamaguchi T, Terashima M, Akasaka T, Hayashi T, Mizuno K, Muramatsu T, Nakamura M, Nakamura S, Saito S, Takano M, Takayama T, Yoshikawa J, Suzuki T. Safety and feasibility of an intravascular optical coherence tomography image wire system in the clinical setting. Am J Cardiol. 2008 Mar 1;101(5):562-7. doi: 10.1016/j.amjcard.2007.09.116. Epub 2008 Jan 10. PMID 18307999
- [Result] Prati F, Cera M, Ramazzotti V, Imola F, Giudice R, Albertucci M. Safety and feasibility of a new non-occlusive technique for facilitated intracoronary optical coherence tomography (OCT) acquisition in various clinical and anatomical scenarios. EuroIntervention. 2007 Nov;3(3):365-70. doi: 10.4244/eijv3i3a66. PMID 19737719
- [Derived] Lee SW, Lam SC, Tam FC, Chan KK, Shea CP, Kong SL, Wong AY, Yung A, Zhang LW, Tse HF, Wu KK, Chan R, Haude M, Mehran R, Mintz GS, Maehara A. Evaluation of Early Healing Profile and Neointimal Transformation Over 24 Months Using Longitudinal Sequential Optical Coherence Tomography Assessments and 3-Year Clinical Results of the New Dual-Therapy Endothelial Progenitor Cell Capturing Sirolimus-Eluting Combo Stent: The EGO-Combo Study. Circ Cardiovasc Interv. 2016 Jul;9(7):e003469. doi: 10.1161/CIRCINTERVENTIONS.115.003469. PMID 27418609